CLINICAL TRIAL: NCT02207179
Title: Breast Cancer Margin Delineation Using Polarization Subtraction Imaging Technology: An Ex-vivo Pilot Study of Real-time Breast Margin Imaging in Women Undergoing Breast Conservation Surgery for Early Stage Breast Cancer
Brief Title: Breast Cancer Margin Delineation Using Polarization Subtraction Imaging Technology
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LumaMed (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM010
Record Dates: First submitted 2014-03-25; First posted 2014-08-04 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Intraoperative; Cancer margin; Spectroscopy; Polarization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (No Intervention): LumaScan Image Guided Surgery
  Interventions: Device: LumaScan Image Guided Surgery

INTERVENTIONS:
Device: LumaScan Image Guided Surgery

SUMMARY:
This study will evaluate LumaScan, an innovative polarization microscope for real time, intraoperative imaging and evaluation of the surface of excised tissue excised during Breast Conservation Surgery (BCS) for non invasive and invasive breast cancer. The investigators hypothesis is that LumaScan will be comparable for cancer detection to conventional histopathologic evaluation of the same areas of breast tissue. The real time, intraoperative images provided by LumaScan will help improve BCS and lessen the need for BCS re-excision surgeries which can lead to higher cost, poor cosmetic outcomes, reduced survival rates, and loss of confidence in the tissue conservation surgery procedure.

DETAILED DESCRIPTION:
LumaScan is an innovative polarization microscope that uses Polarization Subtraction Imaging (PSI) technology to provide real time, intra operative, digital images of the surface of tissue removed during BCS for breast cancer. PSI uses polarized visible light for optical sectioning and geometric imaging of the superficial layers of the surgically removed tissue while rejecting surface scatter and light from deeper layers. By rejecting light from deeper tissues PSI is able to exclusively focus on the superficial tissue layers. This also results in higher resolution images than are possible with standard optical imaging. PSI is used in both reflectance and fluorescence modes. Reflectance detects morphologic abnormalities that occur in tumor progression such as increased nuclear density, angiogenesis, cellular infiltration and crowding while fluorescence detects early biochemical changes.

To enhance the contrast of tumor at the margins the investigators will use Methylene blue (MB), a dye that has been commonly used in breast surgery for mapping sentinel lymph nodes. MB can be administered peritumorally and is quickly taken up by cells in only a few minutes of exposure and its presence does not interfere with or preclude later histopathology on the same tissue specimen. A tumor specimen may also be dipped in MB post-excision to achieve tumor margin contrast enhancement and not interfere with pathologic assessment.

Previous research using PSI technology has demonstrated the value of PSI in mapping tumor boundaries of breast cancer in excised tissue specimens and in non-melanoma skin cancers and these boundaries in side by side comparisons correlate well with those marked by a pathologist on representative sections prepared using standard H&E staining procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Women referred for breast conservation surgery following a diagnosis of invasive or in situ carcinoma of the breast by histopathology or women referred for lumpectomy due to a benign (fibroadenoma or papilloma) or high risk breast lesion(Atypical ductal hyperplasia, atypical lobular hyperplasia, lobular carcinoma in-situ, atypical papilloma).
2. 18 years of age or older.
3. Able to read or understand and give informed consent.

Exclusion Criteria:

1. Patients undergoing neo-adjuvant systemic therapy.
2. Previous breast cancer and /or radiation in the operated breast.
3. Implants in the operated breast.
4. Pregnant or Lactating.
5. History of photosensitizing disease (porphyria, lupus etc.) or of allergy to methylene blue dye.
6. Recent use of photosensitizing agents such as fluoroquinolones and retinoids or patients undergoing phototherapy.
7. Participation in any other intraoperative margin assessment protocol that would affect data acquisition.
8. Subareolar location (cancer is directly and completely under the nipple/areolar complex) of breast abnormality.
9. Patients for whom English is not their native language

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Tumor areas shown on LumaScan images are the same as those shown on subsequent en-face pathology images. | From day of surgery until receipt of pathology results (upto 2 weeks)
  Quantitative metrics (e.g. size or area of tumor found between the two images) will be used to to compare en-face pathology and corresponding LumaScan images from excised breast tissue margins.

SECONDARY OUTCOMES:
Pathologist interpretation of LumaScan images (blinded) are similar to those of histopathology images. | From day of surgery until receipt of pathology results (upto 2 weeks)
  The Pathologists will be asked to interpret LumaScan images and corresponding histopathology images. The images will be randomly presented to the Pathologist in order to be blinded to each.
Surgeons interpretation of LumaScan images (blinded) are similar to those of histopathology images. | From day of surgery until receipt of pathology results (upto 2 weeks)
  To correlate and determine the surgeons blinded interpretation of the LumaScan images, digital photographs vs. the final pathologic outcomes (post image acquisition)
Time for each margin and bi-valved image acquisition in the operating room | Duration of surgery (upto 3 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Lee G Wilke, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States